CLINICAL TRIAL: NCT02868294
Title: Preventive Fixation of Lower Limbs in Osteogenesis Imperfecta (Brittle Bone Disease) With the Highlight of the Fassier-Duval
Acronym: Fassier-Duval
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-06; 2011-A00437-34 (Registry Identifier: IDRCB); RC12_3016 (Other: Assistance Publique Hôpitaux de Marseille)
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Brittle Bone Disease
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient receiving the Fassier-Duval Nail (Experimental): Implementation of a telescopic system intramedullary
  Interventions: Device: Fassier-Duval Nail

INTERVENTIONS:
Device: Fassier-Duval Nail — Implementation of a telescopic system intramedullary

SUMMARY:
Osteogenesis imperfecta (or brittle bone disease) is a rare genetic disease characterized by fragile bone and a low mass ossue, secondary to abnormal collagen synthesis. This is a real congenital osteoporosis. The prevalence of the disease is not known precisely, but it is 1 in 10000 at 20000. There are many forms of osteogenesis imperfecta to classify patients with symptomatology minor to the patients with lethal form during the neonatal period. The main symptoms are dominated by fractures and bone deformities, particularly in the lower limbs. Bisphosphonate medication is used for over 10 years to reduce the number of fractures. However the long-term effects are not known to date, not allowing even to establish proof of the benefit risk. Thus unable to process all of these patients and over a long time, these drug treatment leaves much therapeutic solutions to surgery. The goal of surgery is to treat fractures, treat bone deformities and prevent fractures future. In the long bones of the limbs, the only effective techniques are intramedullary nailing. The majority of realized nailing nailing are either sliding or telescopic enabling having a reinforced bone of an intramedullary osteosynthesis material over its entire length during the period of bone growth. It has been shown that the technique of the sliding nailing was inexpensive but reliable especially before the age of 5 years. After that age, all are telescopic nailing nailing. The first telescopic nail described is the Bailey-Dubow nail still widely used in France. However, the number of complications relating to its use is important. Thus, there are 8% of disunity equipment and 33 to 72% of the nail migration forcing him to change one or more times during growth. A new nail presented at the French orthopedic company in 2005 and Fassier Duval reported a much lower complication rate because the rate of nail migration is only 9%, without opening the knee joint, which is not possible with the highlight of Bailey-Dubow.

It is proposed to conduct a prospective series of 10 nailing the lower extremities with this nail Fassier-Duval in patients with osteogenesis imperfecta and compare the results with a series of patients already treated with Bailey-Dubow nails in order to highlight the advantages and disadvantages of using of such a nail.

ELIGIBILITY:
Inclusion Criteria:

* Minor Patient, male or female patients with osteogenesis imperfecta
* Patients who were operated on for intramedullary nailing of the femur or tibia by a nail-Bailey Dubow or sliding nailing between 1996 and 2010
* Patients with surgical management of the disease was performed in the orthopedic surgery department of the Assistance Publique Hôpitaux de Marseille

Exclusion Criteria:

* Non patients with osteogenesis imperfecta
* Major patients
* Patients who have never had nailing of the femur or tibia by a nail-Bailey Dubow or sliding nailing

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2011-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Assessment by radiography intraosseous migration rate | 72 months
  Measure the distance between the end of a nail with the visible boundaries of the epiphysis and the growth of cartilage.

CONTACTS AND LOCATIONS:
Overall Officials: Franck LAUNAY, PU-PH, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France